CLINICAL TRIAL: NCT07331870
Title: Performance Evaluation of DIY Digital Visual Acuity Test
Acronym: CI01-2022
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ojenforeningen (Other)
Collaborators: Veranex Switzerland SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Ojenforeningen
Record Dates: First submitted 2025-11-21; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Visual Acuity
Keywords: Visual acuity; ETDRS evaluation; Radner test; software based Visual acuity test

STUDY DESIGN:
Masking Description: No making applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Comparaison to standard of Care (Experimental): The measurements performed with the investigational device are compared to the standard of care (ETDRS and Radner test)
  Interventions: Device: Comparaison of the investigation device measurement with standard of Care

INTERVENTIONS:
Device: Comparaison of the investigation device measurement with standard of Care — The patient Visual acuity is measured with the investigational device, the ETDRS method, the radner test and the results are compared.

SUMMARY:
This study aims to verify the accuracy of a new Digital Visual Acuity test. The test results obtained with the support of the device will be compared to the current standard of care related to visual acuity testing.

DETAILED DESCRIPTION:
The investigational device is a software-based application for computers and tablets that enables individuals without professional training to self-assess their near and distance visual acuity. It is a low-risk device and represents an evolution of an already marketed product. The device is intended to support ongoing monitoring for patients with conditions that may affect visual acuity, helping track changes over time. It is not designed to replace a comprehensive eye examination performed by a qualified eye-care professional. For this study, the advanced version of the application will be used.

The study population will include adults with normal, subnormal, and low vision to ensure validation of the test across the full range of visual acuity levels. Participants will include patients attending the Eye Department for treatment of various ocular conditions (low-vision group), as well as patients' spouses and department staff (subnormal and normal vision groups). All participants must be able to make independent judgments. Before participation, each individual will receive information about the study procedures, including the nature of the intervention and their right to withdraw at any time.

The device does not require specialized training. Users will receive a brief initial orientation on how to operate the application. For the home self-test, users will complete the assessment independently and without assistance to evaluate the device's usability and support autonomous testing.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older.
* Subjects must be able to understand and perform the test.
* Subject must have corrected vison (i.e. wearing glasses)

Exclusion Criteria:

* Subjects not able to understand the implications of participating in a scientific study.
* Subjects not legally independent.
* Subjects not able to perform the test.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2025-11-15 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
Agreement of Digital Visual Acuity Test Scores With ETDRS (Distance) and Radner (Near) Visual Acuity Scores | up to 90 days
  Difference and agreement between visual acuity scores obtained using the DIY Digital Visual Acuity Test and scores obtained using the ETDRS chart for distance vision and the Radner chart for near vision, measured in logMAR units.
Repeatability of Visual Acuity Measurements Obtained With the DIY Digital Visual Acuity Test Compared With ETDRS (Distance) and Radner (Near) Charts | up to 90 days
  Within-subject repeatability of visual acuity measurements, expressed in logMAR units, across repeated use of the DIY Digital Visual Acuity Test compared with repeated measurements obtained using ETDRS charts for distance vision and Radner charts for near vision.

CONTACTS AND LOCATIONS:
Overall Officials: Lisbeth Sandfeld, PhD MD, Principal Investigator — Zealand University Hospital, Roskilde, Denmark
Locations (1):
- Eye Dept., Zealand University Hospital, Roskilde, Denmark, Denmark

IPD SHARING:
Plan to Share IPD: No
The current consent obtained by subjects to process their data does not include sharing their data in any form beyond this clinical trial.